CLINICAL TRIAL: NCT01891227
Title: Capecitabine in Combination With Bendamustine in Women With Pretreated Locally Advanced or Metastatic Her2-negative Breast Cancer, a Phase II Trial
Brief Title: Capecitabine + Bendamustine in Women With Pretreated Locally Advanced or Metastatic Her2-negative Breast Cancer
Acronym: MBC-6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_MBC-6
Record Dates: First submitted 2013-06-27; First posted 2013-07-03 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: Bendamustine; Capecitabine; Pretreated; Her2 negative; Advanced breast cancer; Metastatic breast cancer; Anthracycline pretreatment; Taxane pretreatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine and Bendamustine (Experimental): Capecitabine will be dosed at 1000mg/m2 twice daily for 14 days, followed by a 7-day rest period for a total cycle time of 21 days (until disease progression or unacceptable toxic effects).
  Bendamustine 80mg/m2 will be administered on day 1 and 8 of a three week cycle (for a maximum of eight cycles).
  Eligible patients will receive capecitabine in combination with bendamustine for a maximum of eight cycles and afterwards capecitabine mono will be continued until disease progression or unacceptable toxic effects. Safety assessments will be conducted in 3-weekly intervals; efficacy assessments will be conducted every 9 weeks.
  Interventions: Drug: Capecitabine; Drug: Bendamustine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be dosed at 1000mg/m2 twice daily for 14 days, followed by a 7-day rest period for a total cycle time of 21 days (until disease progression or unacceptable toxic effects).
  Other Names: Xeloda
Drug: Bendamustine — Bendamustine 80mg/m2 will be administered on day 1 and 8 of a three week cycle (for a maximum of eight cycles).
  Other Names: Levact

SUMMARY:
Patients with pretreated, Her2-negative, advanced breast cancer will receive chemotherapy with capecitabine and bendamustine for a maximum of eight cycles and afterwards capecitabine alone until disease progression or unacceptable toxic effects. Safety assessments will be conducted in 3-weekly intervals, efficacy assessments (CT or MRI) will be conducted every 9 weeks.

Aim of this study is to determine whether treatment with capecitabine in combination with bendamustine is efficacious and safe.

DETAILED DESCRIPTION:
40 eligible patients will be enrolled. A two-stage design efficacy and safety of bendamustine and capecitabine will be evaluated following recruitment of the first 20 patients. Upon favorable results a further 20 patients will be recruited to reach the target population of 40 evaluable patients.

Pretreatment for eligible patients must include anthracyclines and/or taxanes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Female patients, age ≥ 18 years (women of childbearing potential must have a negative pregnancy test at screening and must use effective contraception)
* Advanced or metastatic Her2-negative breast cancer, histologically confirmed
* At least one measurable lesion according to RECIST criteria (Version 1.1)
* Documented disease progression
* Patients with progression after anthracycline and/or taxane treatment(palliative or adjuvant)
* Life expectancy of at least 12 weeks
* Performance status 0-2
* Hematologic:

  * ANC (absolute neutrophil count) ≥ 1.5 x 109/L
  * Hemoglobin ≥ 9 g/dL
  * Platelets ≥ 100 x 109/L
* Liver Function:

  * Albumin ≥ 2.5 g/dL
  * Serum bilirubin ≤ 2 mg/dL
  * AST (Aspartate aminotransferase) and ALT (Alanine aminotransferase) ≤ 3 x ULN (Upper limit of Normal) without liver metastases

    * 5 x ULN if documented liver metastases
* Renal Function:
* Serum Creatinine ≤ 1.5 mg/dL OR Calculated Creatinine Clearance ≥ 40 mL/min

Exclusion Criteria:

* Pregnant or lactating women
* Serious medical or psychiatric disorders that would interfere with the patient's safety or informed consent
* Radiation of the target lesion within the last 4 weeks
* Active bacterial, viral or fungal infection
* Patients with clinically apparent brain metastases
* Known Positivity for HIV
* Positivity for Hepatitis B or C
* History of other malignancy; patients who have been disease-free for 5 years or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Concurrent cancer therapy (chemotherapy, immunotherapy, antihormonal or biologic therapy) or concurrent treatment with an investigational drug
* Antihormonal therapy must have been discontinued prior to start of treatment (if possible at least 3 weeks before)
* Known hypersensitivity to the study drugs capecitabine and bendamustine or their excipients
* Pretreatment with capecitabine (pretreatment with infusional 5-FU (Fluorouracil) in the adjuvant or neoadjuvant setting is allowed) or bendamustine
* Treatment with sorivudine or derivates e.g. brivudin (Mevir©) within the last 4 weeks before and during study treatment with capecitabine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08-09 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of capecitabine + bendamustine combination regimen | At baseline + every 9 weeks until progression + at end of study treatment; expected study duration 3 years
  Overall response rates (complete or partial response, determined by radiologic evaluation according to Response Evaluation Criteria in Solid Tumors - RECIST (Response Evaluation Criteria In Solid Tumors) Version 1.1) The study will be stopped after 20 patients if there are fewer than four subjects with an overall response of CR (complete response) or PR (partial response). If there are at least four responses an additional 20 subjects will be enrolled and treated till a maximum of 40 subjects. The regimen is concluded to be effective if 13 or more responses out of 40 are observed at the end of the trial.
  The last patient is expected to enter the study in Q1 2015, following a 24 month recruitment period. Last Subject Last Visit will be at final staging after end of treatment of last patient. Follow-up after Last Subject Last Visit will be conducted according to local standard of care thereafter, and is not part of study procedures.

SECONDARY OUTCOMES:
Safety profile of a combination with capecitabine and bendamustine | From treatment start until 28 days after last study treatment; expected study duration 3 years
  To determine the safety profile of a combination with capecitabine and bendamustine in terms of qualitative and quantitative toxicities from first study treatment dose until completion of study treatment due to progression or for any other reason. All safety analyses will be based on the safety population, defined as subjects who received at least one dose of the study medication and have at least one post-treatment safety assessment available. The safety population will be used for all safety and tolerability analyses including demographic data, vital signs, laboratory data and adverse events.
Clinical benefit | Baseline + every 9 weeks until progression + at end of study treatment; expected study duration 3 years
  CR, PR or stable disease for at least 24 weeks
Progression free survival | Baseline + every 9 weeks until progression; expected study duration 3 years
Overall survival | During complete study treatment, after study treatment every 3 months until end of complete study; expected study duration 3 years
  explorative, from treatment start until death from any cause
Quality of life | Baseline + every 9 weeks until progression + at end of study treatment; expected study duration 3 years
  To evaluate Quality of Life (QoL) status within the study population using the EORTC (European Organisation for Research and Treatment of Cancer) QLQ (Quality-of-life-questionnaire)-C30 standard questionnaire and the BR23 module (module for breast cancer patients)
Predefined subgroup analysis in terms of response | Baseline + every 9 weeks until progression + at end of study treatment+every 3 months after end of treatment until end of study; expected study duration 3 years
  Predefined subgroup analysis of triple-negative patients and hormone receptor positive patients in terms of response

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, Prof.Dr., Principal Investigator — Universitätsklinik für Innere Medizin III, Salzburg
Locations (8):
- Austria (8):
  - Hämatologie und Onkologie/Interne E, LKH Feldkirch, Feldkirch
  - Universitätsklinik f. Frauenheilkunde und Geburtshilfe, Klin. Abt. f. Gynäkologie, Graz
  - Universitätsklinik f. Innere Medizin, Klin.Abt. f. Onkologie, Graz
  - Univ.-Klinik f. Frauenheilkunde; Klinische Abt. f. Gynäkologie u. Geburtshilfe, Innsbruck
  - KH Barmh. Schwestern Linz, Innere Medizin I Hämatologie/Onkologie, Linz
  - Kepler Universitätsklinikum, Med Campus III, Klinik f. Interne 3 - Schwerpunkt Hämatologie u. Onkologie, Linz
  - Universitätsklinik für Innere Medizin III, Salzburg
  - Landeskrankenhaus Steyr, Interne Medizin II, Steyr

REFERENCES:
- [Derived] Rinnerthaler G, Gampenrieder SP, Petzer A, Hubalek M, Petru E, Sandholzer M, Andel J, Balic M, Melchardt T, Hauser-Kronberger C, Schmitt CA, Ulmer H, Greil R. Capecitabine in combination with bendamustine in pretreated women with HER2-negative metastatic breast cancer: results of a phase II trial (AGMT MBC-6). Ther Adv Med Oncol. 2021 Oct 19;13:17588359211042301. doi: 10.1177/17588359211042301. eCollection 2021. PMID 34691243